CLINICAL TRIAL: NCT02340429
Title: The Impact of Using a Video Otoscope on Parents' Satisfaction in Pediatric Ear Examination: A Prospective Randomized Controlled Study:
Brief Title: Using a Video Otoscope in Pediatric Ear Examination: A Prospective Randomized Controlled Study:
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ziv Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: ZIV 0094-14
Record Dates: First submitted 2015-01-13; First posted 2015-01-16 (Estimated); Last update posted 2015-07-14 (Estimated); Status verified 2015-01

CONDITIONS: Parental Satisfaction of Using Video Otoscopy in Pediatric Emergency Room

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- video otoscopy (Experimental): children under 18y admitted to the pediatric emergency room for any reason, will undergo video otoscopy
  Interventions: Device: DE500 Digital Video Otoscope
- standard otoscopy (No Intervention): children under 18y admitted to the pediatric emergency room for any reason, undergoing routine otoscopy

INTERVENTIONS:
Device: DE500 Digital Video Otoscope
  Arms: video otoscopy

SUMMARY:
Medical care today is moving towards patient centered care (PC) and patient empowerment (PE), both in practice and in medical staff training . Applying this methodology enhances patient autonomy in the clinical setting and allows shared decision making.

Current mobile and video technology enables the caregiver(clinician) to share visual data with the patient, making him or her a more active participant in the medical procedure. It has been shown that higher patient satisfaction rate regarding the patient/physician encounter, has a positive effect on medical procedure outcome and patient compliance.

Patient centered care and Patient Empowerment benefits are maximized using the proper tools. One such tool is the video otoscope. In this study we apply the PC/PE approach of medical care and introduce video otoscopy in the setting of a pediatric emergency room. We use an affordable (~300$), FDA approved, High Res. video otoscope. (DE500 Digital Video Otoscope,Firefly global Inc.) Patients will be randomized upon admission into two groups: video otoscopy and standard otoscopy. Upon discharge from the pediatric ER, parents will be asked to answer a short questionnaire regarding their satisfaction with the ER visit and the otoscopic examination.

We aim to study the impact of affordable, high res. video otoscopy, on the general satisfaction of parents from their emergency room experience, vs their experience when undergoing a regular otoscopic examination.

Inclusion criteria: children under 18y admitted to the pediatric ER for any reason, undergoing routine otoscopy, who's parents have signed an informed consent.

Exclusion criteria: no parental informed consent,lake of compliance or inability to perform otoscopy.

Number of participants: 60 (30 in each group) Study start: January 2015 Study ends:January 2016 Study location: Ziv medical center, Zefat Israel

ELIGIBILITY:
Inclusion Criteria:

* Children under 18y admitted to the pediatric ER for any reason, undergoing routine otoscopy, who's parents have signed an informed consent.

Exclusion Criteria:

* no parental informed consent, lack of compliance or inability to perform otoscopy.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2015-01; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
parental satisfaction questionnaire | 1 year